CLINICAL TRIAL: NCT01086631
Title: Rituximab for Autoimmune Retinopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100040; 10-EI-0040
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-07-08

CONDITIONS: Autoimmune Disease
Keywords: Autoimmune Retinopathy; RITUXAN; Rituximab; Immunosuppression
MeSH Terms: conditions — Autoimmune Diseases | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
Background:

* Autoimmune retinopathy (AIR) is an inflammatory condition in which the patient s own immune system is attacking his or her eyes and causing vision loss. Patients with AIR are generally treated with immunosuppressive agents to treat the eye inflammation; however, the standard treatment for this disease is still being developed.
* Rituximab, an immunosuppressive agent, is a monoclonal antibody that is directed against a part of the immune system that may be an important cause of AIR. Rituximab is approved for the treatment of non-Hodgkin s lymphoma and rheumatoid arthritis, but is not approved for the treatment of AIR. Researchers are interested in determining whether rituximab may be used to treat AIR.

Objectives:

- To to investigate the safety, tolerability and possible efficacy of rituximab as a treatment for AIR.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with AIR and have visual acuity of 20/200 or better in at least one eye.

Design:

* Before the start of the study, participants will be screened with a medical history, immunization records, a series of eye examinations, a chest X-ray, an electrocardiogram, and blood tests.
* Participants will receive a maximum of two cycles of rituximab during the 18-month study. Each cycle will involve two separate intravenous infusions of rituximab given 2 weeks apart.
* Participants will return to the clinic 6 weeks after the first cycle of rituximab for a safety visit, which will include a routine eye and physical examinations. They will also provide blood and other samples for study.
* After the safety visit, participants will return every 3 months for follow-up visits.
* At the 6-month visit, participants who have successfully or partially responded to rituximab will receive another cycle of treatment. Those who do not respond will not receive another cycle, but will continue to be monitored until the end of the study.

DETAILED DESCRIPTION:
Objective:

Autoimmune retinopathy (AIR) is an ophthalmic disorder in which autoantibodies damage the retina and its components, causing progressive vision loss. AIR has no established treatment, but systemic immunosuppression has shown favorable responses. Rituximab is an immunosuppressive agent which binds specifically to B lymphocytes. The objective of this study is to investigate the safety of rituximab as an effective treatment for AIR.

Study Population:

Five participants with AIR and visual acuity of 20/200 or better in at least one eye will receive rituximab. AIR must be confirmed by immunohistochemical demonstration of serum anti-retinal antibodies on normal, unfixed, frozen rhesus monkey or human retinas, as well as visual field and electroretinography (ERG) changes. Up to seven participants may be enrolled, in order to obtain the five participants to be included in the analysis if participants withdraw prior to receiving rituximab.

Design:

The study duration is 18 months. Rituximab is administered as a cycle consisting of two separate rituximab infusions of 1,000 mg each, two weeks apart. Participants will receive their first rituximab cycle at baseline and evaluated for a second cycle six months later. Treatment success is defined as experiencing a greater than a 25% improvement in ERG response amplitudes or greater than a 3 decibel (dB) improvement in mean deviation on Humphrey Field Analyzer [HFA (30-2)] or improvement in threshold values greater than 0.5 log in existing scotomas or greater than 25% improvement in the area of scotomas on Goldmann Visual Field (GVF) assessment as compared with baseline. As a result, participants could receive a maximum of two cycles in this study. Participants will return to the clinic 6 weeks and 3 months after their first infusion of each cycle for a safety visit. Study visits will continue every three months for the study duration.

Outcome Measures:

The primary outcome is the number of participants who meet the definition of treatment success within six months from baseline. Secondary efficacy outcomes include changes in visual acuity, the number of treatment successes at 9 and 12 months, the number of partial responders at 6, 9 and 12 months, changes in ERG or visual field as demonstrated by the HFA (30-2) or GVF, changes in optical coherence tomography (OCT), changes in fluorescein angiography (FA), changes in serum anti-retinal autoantibody or anti-retinal antibody staining, changes in color vision, positive visual symptoms or nyctalopia and changes in the participants quality-of-life as assessed by the NEI visual function questionnaire. For participants with greater than or equal to 2 ERG measurements available prior to enrollment, an attempt will be made to compare the rate of decline pre-study period to the rate of decline post-enrollment period. Safety outcomes include the number and severity of systemic and ocular toxicities, adverse events, and infections and the proportion of participants with a loss of greater than or equal to 15 ETDRS letter score.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participant must be 18 years of age or older.

Participant must understand and sign the protocol s informed consent document.

Participant must be willing to comply with the study procedures and expected to be able to return for all study visits.

Participant must have a diagnosis of AIR according to the features listed below.

Participants must have demonstrated evidence of anti-retinal antibodies as noted in criterion a and one or more of the clinical manifestations listed in either criterion b or c in order to be considered eligible.

1. Serologic or immunohistochemical demonstration of serum anti-retinal antibodies (on normal, unfixed, frozen rhesus monkey or human retinas.
2. Visual field changes

i. Defects in visual fields [on HFA (30-2) or GVF]

ii. Enlarged blind spot

c. ERG changes

i. Abnormal amplitudes

ii. Prolonged implicit times.

Participant must have visual acuity of 20/200 or better in at least one eye.

Participant must have normal renal function, liver function and blood cell counts, OR has mild abnormalities and is cleared for enrollment by internal medicine.

Participant must agree not to receive any live or live-attenuated vaccinations (e.g., nasal flu vaccine [FluMist ] or Zostavax ) for the duration of the study.

Participant must have clear ocular media and adequate pupillary dilation to permit quality imaging.

Participant must have a negative PPD screening test as defined by the Centers for Disease Control (CDC) unless otherwise cleared by internal medicine (i.e., previously treated for a positive PPD or a history of Bacillus of Calmette and Guerin (BCG) vaccination).

Female participants of childbearing potential must not be pregnant or breast-feeding, must have a negative serum pregnancy test at screening and must be willing to undergo pregnancy tests throughout the study.

Both female participants of childbearing potential* and male participants able to father a child must agree to practice two** forms of adequate contraception throughout the course of the study and for 12 months following the last administration of the investigational product. Acceptable methods of contraception include hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation or vasectomy).

*Childbearing potential must be determined

**Participants with a hysterectomy or vasectomy (or who have a partner with a hysterectomy or vasectomy) are exempt from using two methods of contraception. However, participants with a tubal ligation (or male participants who have a female partner with a tubal ligation) are not exempt, and are required to practice another acceptable method of contraception.

EXCLUSION CRITERIA:

Participant received other biologic agents (e.g., infliximab, daclizumab or adalimumab) within three months prior to study enrollment.

Participant is receiving more than two immunosuppressive agents or experienced a change in his/her AIR immunosuppressive medication regimen within the two months prior to enrollment.

Participant received intraocular or periocular steroid injections within two months prior to study enrollment.

Participant has a significant active infection (an infection requiring treatment as determined by the medical team) or a history of chronic or recurrent infections.

Participant is HIV positive or has syphilis.

Participant has a history of cancer (other than a non-melanoma skin cancer or non-Hodgkin s lymphoma [NHL]) diagnosed within the past five years.

Participant has or is a carrier of hepatitis B or C.

Participant has a known hypersensitivity to sodium fluorescein dye.

Participant has congestive heart failure, abnormal cardiac function or significant pulmonary disease.

Participant is participating in another simultaneous investigational product treatment trial.

Participant received a live or live-attenuated vaccine within the previous four weeks prior to study enrollment

Participant had ocular surgery within 60 days prior to study enrollment or is anticipated to require elective intraocular surgery.

Participant has inadequately controlled diabetes.

Participant has a condition that, in the opinion of the investigator, would pose a significant hazard to the participant if the investigational product was initiated.

Participant has any other condition that would be contraindicated to treatment with rituximab or their current immunosuppressive agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01-22; Study Completion 2014-07-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the number of participants who meet the definition of treatment success within six months from baseline.

SECONDARY OUTCOMES:
Changes in visual acuity, number of treatment successes or partial responders, changes in ERG, HFA, OCT or FA, changes in serum antibody staining, changes in color vision, and changes in quality-of-life.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Weinstein JM, Kelman SE, Bresnick GH, Kornguth SE. Paraneoplastic retinopathy associated with antiretinal bipolar cell antibodies in cutaneous malignant melanoma. Ophthalmology. 1994 Jul;101(7):1236-43. doi: 10.1016/s0161-6420(94)31183-3. PMID 8035987
- [Background] Jacobson DM, Thirkill CE, Tipping SJ. A clinical triad to diagnose paraneoplastic retinopathy. Ann Neurol. 1990 Aug;28(2):162-7. doi: 10.1002/ana.410280208. PMID 2171418
- [Background] Weleber RG, Watzke RC, Shults WT, Trzupek KM, Heckenlively JR, Egan RA, Adamus G. Clinical and electrophysiologic characterization of paraneoplastic and autoimmune retinopathies associated with antienolase antibodies. Am J Ophthalmol. 2005 May;139(5):780-94. doi: 10.1016/j.ajo.2004.12.104. PMID 15860281